CLINICAL TRIAL: NCT04028115
Title: Bone Healing During Ninlaro Exposure. An Open Label Phase 2 Single Centre Clinical Trial
Brief Title: Bone Healing During Ninlaro Exposure
Acronym: BONE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Thomas Lund (Other)
Responsible Party: Sponsor-Investigator, Thomas Lund, Pd.D Associate Professor Chief Physician, Odense University Hospital
Organization: Odense University Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HFE-X 18.01
Record Dates: First submitted 2019-07-17; First posted 2019-07-22 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Multiple Myeloma
Keywords: WH 540
MeSH Terms: conditions — Multiple Myeloma | interventions — ixazomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Interventional (Experimental): Patients included in the trial will be treated with Ixazomib 4 mg on day 1, 8, and 15 in a 28-day cycle for up to 24 cycles. In this, study no randomisation will occur. All patients will receive the same treatment.
  Interventions: Drug: Ixazomib

INTERVENTIONS:
Drug: Ixazomib — Scheduled visits: Patients included in the trial will be treated with Ixazomib 4 mg on day 1, 8, and 15 in a 28-day cycle for up to 24 cycles. Patients will be evaluated every 4th week by a medical doctor, prior to initiation of a new cycle of Ixazomib.
  Other Names: Ninlaro

SUMMARY:
The primary purpose of this study is to investigate if treatment with Ixazomib in multiple myeloma (MM) can strengthen the bones, thus making it resilient to future fractures. Ixazomib will be given at a time point when the disease is in a stable phase, decreasing the likelihood that the potential bone anabolic effect will be abrogated by catabolic effect of active MM. In order to be included in the study, the patient must have treatment demanding MM, and the disease must have been brought into at least partial remission with chemotherapy before inclusion. Moreover, the patient must have pathological bone structure on low dose CT due to the pre-existing disease.

DETAILED DESCRIPTION:
The primary purpose of this study is to investigate if treatment with Ixazomib in multiple myeloma (MM) can strengthen the bones, thus making it resilient to future fractures. Ixazomib will be given at a time point when the disease is in a stable phase, decreasing the likelihood that the potential bone anabolic effect will be abrogated by catabolic effect of active MM. In order to be included in the study, the patient must have treatment demanding MM, and the disease must have been brought into at least partial remission with chemotherapy before inclusion. Moreover, the patient must have pathological bone structure on low dose CT due to the pre-existing disease.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic Multiple Myeloma according to the IMWG criteria.
* Detectable osteolysis on low dose CT (at least 5 mm in size).
* Stable disease, defined as no signs of progressive disease for three months without anti myeloma treatment.
* Achieved, partial response or better, during last line of therapy.
* Signed informed consent.
* Age ≥ 18 years.
* Remaining life expectancy ≥ 6 months.
* ECOG performance status 0-2.

Female patients who

* Are postmenopausal for at least 1 year before the screening visit, OR
* Are surgically sterile, OR
* If they are of childbearing potential, agree to practice 2 effective methods of contraception, simultaneously, from the time of signing the informed consent form through 90 days after the last dose of study drug, OR
* Agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence (eg, calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception).

Male patients, even if surgically sterilized (i.e., status post-vasectomy), must agree to one of the following

* Agree to practice effective barrier contraception during the entire study treatment period and through 90 days after the last dose of study drug, OR
* Agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence (eg, calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception).

Exclusion Criteria:

* Treatment with Denosumab within the last 4 weeks.
* Known concurrent malignancy (last five years), excluding skin cancer.
* Known hypersensitivity to Ixazomib.
* Central nervous system involvement.
* Ongoing or active systemic infection, active hepatitis B or C virus infection, or known human immunodeficiency virus (HIV) positive Pregnant or lactating women
* Absolute neutrophil count < 1,000mm3 without growth factor support.
* Platelet count < 75,000/mm3. Platelet transfusions to help patients meet eligibility criteria are not allowed within 3 days before inclusion -Total bilirubin > 1.5 x the upper limit of the normal range.
* Alanine aminotransferase > 3 x upper limit of the normal range.
* Calculated creatinine clearance < 30 mL/min (using the Cockcroft-Gault equation).
* Total bilirubin > 1.5 the upper limit of the normal range (ULN).
* Radiotherapy within 14 days before inclusion.
* Major surgery within 14 days before inclusion.
* Evidence of current uncontrolled cardiovascular conditions, including uncontrolled hypertension, uncontrolled cardiac arrhythmias, uncontrolled congestive heart failure, unstable angina, or myocardial infarction within the past 6 months.
* Systemic treatment with strong CYP3A inducers (rifampin, rifapentine, rifabutin, carbamazepine, phenytoin, phenobarbital) or use of St. John's wort.
* Peripheral neuropathy grade 1 with pain or grade 2.
* Participation in other clinical trials, including those with other investigational agents not included in this trial, within 30 days of the start of this trial and throughout its.
* Known GI disease or GI procedure that could interfere with the oral absorption or tolerance of Ixazomibzomib including difficulty swallowing.
* Infection requiring systemic antibiotic therapy or other serious infection within 14 days before study enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-10-24 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
Healing of osteolytic bone lesions on low dose CT. | from the inclusion in the protocol until the patient has been in the protocol for 24 months or until the patient leaves the protocol if that happens before 24 months
  Healing of osteolytic bone lesions on low dose CT. Healing will be evaluated based on the preexisting lesion on low dose CT required upon inclusion. All lesions will be evaluated individually using the inclusion scanning as reference. Healing will be defined as ≥ 25% reduction in the size of osteolytic lesions (a reduction of at least 2 mm in the longest dimension is required), increased sclerosis in the edge of existing lesions, or healing of existing lesions.

SECONDARY OUTCOMES:
Increased bone formation during Ixazomib treatment in NaF PET. | 3, 12 and 24 months
  Increased bone formation during Ixazomib treatment in NaF PET. Increased bone formation will be evaluated in NaF PET by comparing delta values of SUVmax of the individual lesions. The inclusion scan will be used as reference. NaF PET scan will be conducted 45 (+/-5 minutes) minutes after infusion of the NaF tracer.
Increased bone anabolism during Ixazomib treatment. | 3, 12 and 24 months
  Increased bone anabolism during Ixazomib treatment. The bone anabolic markers bALP, PINP, and OC will be measured at screening and during treatment. The patient will function as his or her own control, using the bone marker levels at inclusion as reference.
Increased bone formation to bone degradation ratio during Ixazomib treatment. | 3, 12 and 24 months
  Increased bone formation to bone degradation ratio during Ixazomib treatment. In addition to the anabolic bone markers; the degradation markers CTX and TRAP5b will also be measured. Again using the levels at inclusion, a ratio of bone formation to bone degradation markers will be calculated. Delta values will be calculated during Ixazomib treatment to investigate if bone remodeling changes toward a more anabolic equilibrium.
Increased bone formation using bone histomorphometric evaluation. | 3, 12 and 24 months
  Increased bone formation using bone histomorphometric evaluation. At inclusion and at predefined selected time points, the patient will have a bone marrow biopsy performed. This biopsy will be stored for later evaluation. Evaluation will be conducted using a slightly modified Masson trichrome staining.
Changes in the patients' mesenchymal stroma cells toward a more osteoblastic state. | 3, 12 and 24 months
  Changes in the patients' mesenchymal stroma cells toward a more osteoblastic state. At inclusion and after three months, the patients will have a bone marrow biopsy performed. Stromal cells will be harvested, characterized by Cluster of Differentiation markers, methylation changes, global mRNA expression, and grown in culture assays to investigate their osteoblastic potential.
Investigate safety and toxicities during Ixazomib treatment. | 2 years
  Investigate safety and toxicities during Ixazomib treatment. Ixazomib has been approved by EMEA in combination with Lenalidomide and Dexamethasone in patients who has relapse of MM after initial therapy. Here, we also wish to give Ixazomib after initial therapy has been completed. However, we wish to give it as monotherapy to patients who do not have active disease. Any toxicity during the study will be registered and graded according to NCI CTCAE version 4 National Cancer Institute Common Terminology Criteria for Adverse Events. (Most recent version can be found at: http://ctep.cancer.gov/protocolDevelopment/electronic_applications/ctc.htm).
Depth of cancer response to Ixazomib treatment. | 2 years
  Depth of cancer response to Ixazomib treatment. Ixazomib has an anti-myeloma effect. During the trial, serum and urine M-component as well as serum free light kappa and lambda chains will be measured. Any upgrading of depth of response will be measured in relation to the status prior to the preexisting disease levels before the last treatment was initiated. In addition, changes in disease status during treatment compared to disease burden at inclusion will also be investigated. Bone marrow examination will be done to verify CR. Response is measured according to the International Myeloma Working Group Uniform Response Criteria (2016) appendix 1.
Adherence to therapy. | 2 years
  Adherence to therapy. Ixazomib will be given for up to 24 cycles or until disease progression (biochemical or symptomatic), see appendix 1 for details, unacceptable toxicities, or withdrawal of consent. In the study we will register time on treatment and reason for discontinuation. As a subpart of this, we will also register time to disease progression during Ixazomib treatment, by calculating from the time when the last treatment was initiated and stopped.
Healing of osteolytic bone lesions on low dose CT. | 3, 12, and 24 months
  Healing of osteolytic bone lesions on low dose CT. Healing will be evaluated based on the preexisting lesion on low dose CT required upon inclusion. All lesions will be evaluated individually using the inclusion scanning as reference. Healing will be defined as ≥ 25% reduction in the size of osteolytic lesions (a reduction of at least 2 mm in the longest dimension is required), increased sclerosis in the edge of existing lesions, or healing of existing lesions.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Lund, Ph.D., MD, Principal Investigator — Odense University Hospital
Locations (1):
- Odense University Hospital, Odense, Denmark

REFERENCES:
- [Derived] Levring MB, Diaz-delCastillo M, Gundesen MT, Cedile O, Andersen CW, Nielsen AL, Moller HEH, Vinholt PJ, Asmussen JT, Kristensen IB, Nyvold CG, Kassem M, Abildgaard N, Andersen TL, Lund T. Ixazomib treatment has a dual effect on bone remodeling in patients with multiple myeloma: follow-up results from a phase 2 clinical study. Bone. 2025 Dec;201:117660. doi: 10.1016/j.bone.2025.117660. Epub 2025 Sep 23. PMID 40998041